CLINICAL TRIAL: NCT06545409
Title: Use of Serratus Posterior Superior Intercostal Plane Block in Robotic-Assisted Thoracoscopic Surgery for Thymectomy: A Randomized Controlled Trial
Brief Title: Serratus Posterior Superior Intercostal Plane Block in Robotic-Assisted Thymectomy
Acronym: SPRATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6729
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: RATS Surgery; Thymectomy; Locoregional Anesthesia; Postoperative Pain Management; Serratus Posterior Superior Intercostal Plane Block; Robotic-Assisted Thoracoscopic Surgery
Keywords: SPSIP; RATS Thymectomy; Thymoma
MeSH Terms: conditions — Thymoma | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIP group (Experimental): Patients in this group will be treated with the Serratus Posterior Superior Intercostal Plane Block, administered under ultrasound guidance 15 minutes before surgery in the operating room. The block will be performed by administering 30 ml of 0.25% bupivacaine.
  Interventions: Procedure: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block performed with 0.25% bupivacaine
- Placebo group (Placebo Comparator): Patients in this group will be treated with the Serratus Posterior Superior Intercostal Plane Block, administered under ultrasound guidance 15 minutes before surgery in the operating room. The block will be performed using 30 ml of a placebo solution without an active ingredient (0.9% NaCl)
  Interventions: Procedure: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block performed with a placebo solution (0.9% NaCl)

INTERVENTIONS:
Procedure: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block performed with 0.25% bupivacaine — While the patient is in the prone or the sitting position, a high-frequency linear transducer is placed transversely at the level of the scapular spine, visualizing the upper medial border of the scapula, trapezius muscle, rhomboid major, serratus posterior superior muscle, and the second and third ribs. Next, the transducer is rotated to obtain an oblique view, including the upper medial border of the scapula. The needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs to reach the fascial plane between the serratus posterior superior muscle and intercostal muscles using the in-plane technique. Once the needle contacts the rib, 30 mL of 0.25% bupivacaine is administered superficially to the intercostal muscle.
  Other Names: SPSIP Block with 0.25% bupivacaine
  Arms: SPSIP group
Procedure: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block performed with a placebo solution (0.9% NaCl) — While the patient is in the prone or the sitting position, a high-frequency linear transducer is placed transversely at the level of the scapular spine, visualizing the upper medial border of the scapula, trapezius muscle, rhomboid major, serratus posterior superior muscle, and the second and third ribs. Next, the transducer is rotated to obtain an oblique view, including the upper medial border of the scapula. The needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs to reach the fascial plane between the serratus posterior superior muscle and intercostal muscles using the in-plane technique. Once the needle contacts the rib, 30 mL of 0.9% NaCl is administered superficially to the intercostal muscle
  Other Names: SPSIP Block with placebo solution (0.9% NaCl)
  Arms: Placebo group

SUMMARY:
This study aims to assess the effectiveness of the Serratus Posterior Superior Intercostal Plane Block (SPSIP Block) for postoperative pain control, reducing opioid analgesic consumption, minimizing postoperative respiratory complications, and enhancing patient satisfaction (measured using the QoR-15 index) in patients undergoing robotic thymectomy, compared to patients who do not receive the block.

DETAILED DESCRIPTION:
All patients enrolled in the study will receive the SPSIP Block under ultrasound guidance 15 minutes before entering the operating room. The SPSIP Block will be performed by the attending anesthetist (investigator 1), who will use a syringe pre-filled with 30 ml of a solution prepared in advance by another investigator (investigator 2). According to the randomization scheme, the solution in the syringe used for the SPSIP Block will contain either 0.25% bupivacaine for 50% of the cases (SPSIP group) or sterile saline solution (0.9% NaCl) for the remaining 50% of the cases (control group). Postoperatively, data collection will be managed by a third investigator (investigator 3). Neither the investigator 1, the patient, nor the investigator 3 will be informed of the syringe's contents, ensuring the study is conducted blind.

All patients enrolled in the study will receive 1000 mg of paracetamol and 30 mg of ketorolac at the end of the surgery, during skin closure. Additionally, upon arrival in the recovery room, all patients will be connected to a PCA (Patient Controlled Analgesia) pump filled with a solution containing opioids. Patients who have NPRS scores greater than 4 during postoperative pain reassessments, despite PCA use, will be given a rescue analgesic dose of 1000 mg of paracetamol (which can be repeated after 8 hours, up to a maximum of 3000 mg in 24 hours).

Postoperative pain intensity will be assessed by investigator 3 at 0, 2, 6, 12, and 24 hours after the end of surgery using the Numeric Pain Rating Scale (NPRS). Assessments will be conducted both at rest and during coughing. Total opioid and rescue analgesic consumption, incidence of postoperative complications, and length of hospital stay will also be recorded. Twenty-four hours after the surgery, investigator 3 will administer the Quality of Recovery 15 (QoR-15) questionnaire to all patients enrolled in the study. The responses will be used by investigator 3 to calculate the QoR-15 Index, which summarizes the degree of patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by thymoma, thymic hyperplasia, or thymic pathologies (cysts, teratomas) who have given informed consent to the study.

Exclusion Criteria:

* Patients who refuse to participate in the study by not signing the informed consent;
* Patients with myasthenia gravis, severe obesity (BMI > 35), history of OSAS with or without CPAP;
* Patients belonging to ASA classes > 3, according to the system developed by the American Society of Anesthesiologists;
* Patients unable to understand the functioning of the NPR Scale or the PCA device that will be used for postoperative analgesia;
* Patients with allergies to analgesic and/or anesthetic drugs;
* Patients on anticoagulant therapy;
* Patients with a history of chronic pain;
* Patients with an infection at the site where SPSIPB will be performed;
* Patients who have had previous thoracic surgery and/or thoracic trauma with rib fractures on the side of the surgery;
* Patients with chest deformities and/or neuromuscular diseases that interfere with normal ventilatory function.

Additionally, patients whose surgery is intraoperatively converted to sternotomy thymectomy will be excluded post-hoc from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | 0, 2, 6, 12, and 24 hours after the end of the surgical procedure
  The measurement of postoperative pain intensity, assessed using the Numeric Pain Rating Scale (NPRS), a numerical scale that can range from 0 to 10 (where 0 means no pain and 10 corresponds to the worst imaginable pain), in the two study groups.

SECONDARY OUTCOMES:
Total opioid drug consumption | 24 hours after surgery
  The total number of opioid doses administered via a Patient Controlled Analgesia (PCA) device in the first 24 hours after surgery
Consumption of rescue analgesics | 24 hours after surgery
  The total dose of acetaminophen administered upon the patient's request during the first 24 postoperative hours
postoperative respiratory complications | 24 hours after surgery
  The number of any postoperative respiratory complications in the two study groups
postoperative quality of recovery | 24 hours after surgery
  the patient's level of satisfaction measured using the QoR-15 index, a numerical parameter calculated by administering the Quality of Recovery 15 (QoR-15) questionnaire to the patient
Length of Hospital Stay | from the end of the surgical procedure to patient discharge
  the duration of postoperative hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Punzo, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS; Dania Nachira, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico A.Gemelli IRCCs, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CQ, Wang J, Liu FY, Wang W. Robot-assisted thoracoscopic surgery vs. sternotomy for thymectomy: A systematic review and meta-analysis. Front Surg. 2023 Jan 6;9:1048547. doi: 10.3389/fsurg.2022.1048547. eCollection 2022. PMID 36684131
- [Background] Chao YK, Lee JY, Lu HI, Tseng YL, Lee JM, Huang WC. Robot-assisted surgery outperforms video-assisted thoracoscopic surgery for anterior mediastinal disease: a multi-institutional study. J Robot Surg. 2024 Jan 13;18(1):21. doi: 10.1007/s11701-023-01745-1. PMID 38217569
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- [Background] Avci O, Gundogdu O, Balci F, Tekcan MN, Ozbey M. Efficacy of serratus posterior superior intercostal plane block (SPSIPB) on post-operative pain and total analgesic consumption in patients undergoing video-assisted thoracoscopic surgery (VATS): A double-blinded randomised controlled trial. Indian J Anaesth. 2023 Dec;67(12):1116-1122. doi: 10.4103/ija.ija_589_23. Epub 2023 Dec 13. PMID 38343684
- [Result] Shintani Y, Funaki S, Ose N, Kanou T, Fukui E, Kimura K, Minami M. Surgical management of thymic epithelial tumors. Surg Today. 2021 Mar;51(3):331-339. doi: 10.1007/s00595-020-02070-y. Epub 2020 Jul 10. PMID 32647929